CLINICAL TRIAL: NCT04663945
Title: Predictors of Recovery and the App-Facilitated Tele-Rehabilitation (AFTER) Program for COVID Survivors
Brief Title: Predictors of Recovery and the App-Facilitated Tele-Rehabilitation (AFTER) Program for COVID-19 Survivors
Acronym: AFTER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-2415
Record Dates: First submitted 2020-12-08; First posted 2020-12-11 (Actual); Results first posted 2022-11-04 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-10

CONDITIONS: Covid-19; Deconditioning
Keywords: Tele-rehabilitation; High Intensity; Biobehavioral; Activity Self-Monitoring; Physical Functional Performance
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): This group will receive 12 biobehaviorally informed tele-rehabilitation sessions including high-intensity strengthening; sessions will be delivered by a licensed physical therapist. An application ('Platform') will facilitate home exercise program completion outside of the supervised sessions.
  Other: remote controlled exercise plus home exercise
  Treatments: strengthening, balance, functional activities, stretching, breathing, aerobic endurance exercise
  Interventions: Behavioral: Biobehavioral Tele-rehabilitation Sessions
- Control (No Intervention): This group will receive an activity monitor and basic education, but no individualized rehabilitation sessions or biobehavioral training.
  Other: basic education

INTERVENTIONS:
Behavioral: Biobehavioral Tele-rehabilitation Sessions — Biobehavioral tele-rehabilitation sessions
  Arms: Intervention

SUMMARY:
The aim of this study is to investigate the feasibility (safety, adherence) and initial efficacy (physical function and patient reported outcomes) of a multicomponent tele-rehabilitation program during COVID-19 recovery of patients who have been hospitalized due to COVID-19.

DETAILED DESCRIPTION:
The aim of this study is to investigate the feasibility and initial efficacy of a multicomponent tele-rehabilitation program during COVID-19 recovery. The tele-rehabilitation program will include biobehavioral training and high intensity exercise facilitated through an online application ('Platform'). Initial efficacy will be assessed primarily by performance on the 30" Chair Stand Test and secondarily through other physical function tests and patient reported outcome measures.

This study will advance the feasibility of tele-rehabilitation as a more generally useful intervention in patients lacking access (distance, availability, mobility) to standard rehabilitative services and could transform the way in which acute rehabilitation and post-hospital care is delivered for all patients.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed COVID-19, per diagnostic criteria (PCR testing)
2. Hospitalized for at least 24 hours
3. Able to provide informed consent
4. Internet capability to access the platform
5. Community-dwelling prior to hospitalization

Exclusion Criteria:

1. Unstable medical comorbidities that would preclude participation in exercise
2. Receipt of >1 session of outpatient physical therapy
3. Known pregnancy, as the impact on physical function, pulmonary function, and other outcomes will vary well beyond any expected effects of COVID-19
4. Anticipating concurrent additional physical therapy services during study intervention period (12 weeks)

Ages: 35 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2020-12-11 (Actual); Primary Completion 2021-08-12 (Actual); Study Completion 2021-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristine Erlandson, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon written request of the study team and an established data use agreement (DUA) between the University of Colorado Anschutz Medical Campus (UCD-AMC) and the requestor's institution, we will provide a deidentified dataset including a data dictionary. Deidentification of the datasets will be conducted with respect to HIPAA definitions, with add back of variables that express all dates as number of days since a milestone event, enrollment, and a variable storing just the year. For example, the milestone event would be "Day 0" in this case.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The main study results will be posted in ClinicalTrials.gov and will remain there indefinitely. All other study documents and data will be made available within a reasonable time frame following a valid written request.
Access Criteria: Other related study documents will be made available upon reasonable written request

REFERENCES:
- [Derived] Churchill L, Morrow M, Capin JJ, Jolley SE, Hare K, MaWhinney S, Stevens-Lapsley JE, Erlandson KM. Using Wearable Technology to Quantify Physical Activity Recovery: Secondary Report From the AFTER (App-Facilitated Tele-Rehabilitation) Program for COVID-19 Survivors Randomized Study. JMIR Rehabil Assist Technol. 2023 Mar 20;10:e43436. doi: 10.2196/43436. PMID 36939818
- [Derived] Capin JJ, Jolley SE, Morrow M, Connors M, Hare K, MaWhinney S, Nordon-Craft A, Rauzi M, Flynn S, Stevens-Lapsley JE, Erlandson KM. Safety, feasibility and initial efficacy of an app-facilitated telerehabilitation (AFTER) programme for COVID-19 survivors: a pilot randomised study. BMJ Open. 2022 Jul 26;12(7):e061285. doi: 10.1136/bmjopen-2022-061285. PMID 35882451

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 5 participants screen failed after enrolling, prior to starting the study.
Groups:
- Intervention: This group will receive 12 biobehaviorally informed tele-rehabilitation sessions including high-intensity strengthening; sessions will be delivered by a licensed physical therapist. An application ('Platform') will facilitate home exercise program completion outside of the supervised sessions.
  Other: remote controlled exercise plus home exercise
  Treatments: strengthening, balance, functional activities, stretching, breathing, aerobic endurance exercise
  Biobehavioral Tele-rehabilitation Sessions: Biobehavioral tele-rehabilitation sessions
Period: Overall Study
Arm/Group | Intervention | Control
Started | 29 | 15
Week 6 Evaluation | 28 | 13
Week 12 Evaluation | 28 | 12
Completed | 28 | 12
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Population: Demographics data was only reported for participants who completed the Week 6 evaluation.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 28 | 13 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (10) | 54 (10) | 52 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 5 | 18
  Male | 15 | 8 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 6 | 12
  Not Hispanic or Latino | 22 | 7 | 29
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 5 | 1 | 6
  White | 17 | 7 | 24
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 28 | 13 | 41
30 Second Chair Stand Test [Mean (Standard Deviation); unit: Completions] — The test uses a standard height chair and requires the participant to stand up and sit down as many times as possible in 30 seconds. More completions indicate better physical function. To facilitate accuracy of the test over video, the participant will be instructed to count out loud each time he/she stands. Further, the test will also be facilitated by the Platform.
  Completions | 12 (3) | 11 (3) | 12 (3)
Timed Up-and-Go Test (TUG) [Mean (Standard Deviation); unit: seconds] — The TUG test measures the time it takes for a person to rise from a chair, walk 3 meters, turn around, walk back to the chair, and sit down. Participants will complete the TUG test twice and the best time will be used. Faster times indicate better physical function and lower risk of falls.
  seconds | 10 (3) | 9 (3) | 9 (3)
4-Stage Balance Test [Mean (Standard Deviation); unit: scores on a scale] — The 4-stage balance test measures static balance in 4 different positions (narrow base of support, semi-tandem, tandem, and single-leg). The test is facilitated by the Platform; it requires participants to hold each position for up to 10 seconds. If a participant is unable to hold a position for 10 seconds, the next hardest position is not performed. Completing higher levels indicate lesser fall risk and better balance. Total scores range from 0 to 40, with higher scores indicating better outcomes.
  scores on a scale | 37 (5) | 37 (5) | 37 (5)

OUTCOME MEASURES:

1. Primary Outcome: Adherence (Primary Feasibility/Safety Outcome)
Description: Feasibility will be measured by program adherence, defined as the number of sessions attended divided by the total number of prescribed sessions (n=12). Individuals will be considered adherent if they attend at least 75% (n=9) of the total sessions. Adherence will be collected in the intervention group only.
Time Frame: 12 weeks
Population: Adherence was collected in the intervention group only.
Measure: Mean (95% Confidence Interval); unit: % of participants meeting adherence
Arm/Group | Intervention | Control
Number analyzed (Participants) | 28 | 0
% of participants meeting adherence | 93 [77 to 99] |

2. Primary Outcome: Change in 30 Second Chair Stand Test (Primary Efficacy Outcome)
Description: The test uses a standard height chair and requires the participant to stand up and sit down as many times as possible in 30 seconds. More completions indicate better physical function. To facilitate accuracy of the test over video, the participant will be instructed to count out loud each time he/she stands. Further, the test will also be facilitated by the Platform.
Time Frame: Change from Baseline to 6 weeks (primary end point), persisting at 12 weeks
Population: The control group had one participant who did not complete week 12 testing.
Measure: Mean (95% Confidence Interval); unit: Completions
Arm/Group | Intervention | Control
Number analyzed (Participants) | 28 | 13
Completions
  Change at Week 6 | 3.1 [1.7 to 4.5] | 5.0 [3.1 to 6.9]
  Change at Week 12: number analyzed (Participants) | 27 | 12
  Change at Week 12 | 3.2 [1.8 to 4.6] | 5.1 [3.2 to 7.0]

3. Secondary Outcome: System Usability Scale (SUS)
Description: The SUS is a 10-item survey that uses a 5-point Likert scale (Strongly disagree (1) to Strongly agree (5)). Scores range from 0 to 100 and higher scores indicate better usability. The SUS will be collected in the intervention group only.
Time Frame: 6 weeks (primary end point)
Population: SUS was only collected on Intervention Group
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 26 | 0
score on a scale | 72 [61 to 75] |

4. Secondary Outcome: Safety Event Count
Description: The Safety Event Count is the cumulative number of participants who experienced adverse events and severe adverse events counted from baseline to week 12. Events will be categorized by type.
Time Frame: Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 28 | 13
Participants
  Serious Adverse Events | 0 | 1
  Non-Serious Adverse Events | 11 | 9

5. Secondary Outcome: Timed Up-and-Go Test (TUG)
Description: The TUG test measures the time it takes for a person to rise from a chair, walk 3 meters, turn around, walk back to the chair, and sit down. Participants will complete the TUG test twice and the best time will be used. Faster times indicate better physical function and lower risk of falls.
Time Frame: Change from Baseline to 6 weeks (primary end point), persisting at 12 weeks
Population: The control group had one participant who did not complete week 12 testing.
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Intervention | Control
Number analyzed (Participants) | 28 | 13
seconds
  Change at Week 6 | -1.7 [-2.9 to -0.5] | -0.6 [-2.3 to 1.0]
  Change at Week 12: number analyzed (Participants) | 27 | 12
  Change at Week 12 | -1.9 [-3.1 to -0.7] | -0.6 [-2.3 to 1.0]

6. Secondary Outcome: 4-Stage Balance Test
Description: The 4-stage balance test measures static balance in 4 different positions (narrow base of support, semi-tandem, tandem, and single-leg). The test is facilitated by the Platform; it requires participants to hold each position for up to 10 seconds. If a participant is unable to hold a position for 10 seconds, the next hardest position is not performed. Completing higher levels indicate lesser fall risk and better balance. Total scores range from 0 to 40, with higher scores indicating better outcomes.
Time Frame: Change from Baseline to 6 weeks (primary end point), persisting at 12 weeks
Population: The control group had one participant who did not complete week 12 testing.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 28 | 13
score on a scale
  Change at Week 6 | 1.8 [-.01 to 3.6] | 1.6 [-0.9 to 4.1]
  Change at Week 12: number analyzed (Participants) | 27 | 12
  Change at Week 12 | 2.9 [1.1 to 4.7] | 2.7 [0.3 to 5.2]

7. Secondary Outcome: MRC Dyspnea
Description: The MRC dyspnea scale is an interviewer-administered or self-report assessment of the perception of difficulty breathing during five different tasks. Participants respond either yes or no to each task. Score is the sum of the number of Yes answers, 0-5. Higher numbers indicate more difficulty breathing
Time Frame: Change from Baseline to 6 weeks (primary end point), persisting at 12 weeks
Population: The control group had one participant who did not complete week 12 testing.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 28 | 13
score on a scale
  Change at Week 6 | -1.3 [-2.0 to -0.7] | -1.2 [-2.1 to -0.3]
  Change at Week 12: number analyzed (Participants) | 28 | 12
  Change at Week 12 | -1.5 [-2.1 to -0.8] | -1.4 [-2.2 to -0.5]

8. Secondary Outcome: Activities-Specific Balance Confidence (ABC) Scale
Description: The ABC Scale is a 16-item self-report measure of balance confidence in performing activities without losing balance or experiencing a sense of unsteadiness. Score range: 0-100. Higher scores indicate higher confidence in performing activities without losing balance.
Time Frame: Change from Baseline to 6 weeks (primary end point), persisting at 12 weeks
Population: The control group had one participant who did not complete week 12 testing.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 28 | 13
score on a scale
  Change at Week 6 | 7.1 [-0.2 to 14.3] | 11.3 [1.6 to 21.1]
  Change at Week 12: number analyzed (Participants) | 28 | 12
  Change at Week 12 | 10.0 [2.7 to 17.3] | 14.2 [4.5 to 24.0]

9. Secondary Outcome: Three-Item Loneliness Scale
Description: This scale has three items and a simplified set of response categories that is designed to measure overall loneliness. Score range: 3-9. Higher scores indicate higher loneliness.
Time Frame: Change from Baseline to 6 weeks (primary end point), persisting at 12 weeks
Population: The control group had one participant who did not complete week 12 testing.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 28 | 13
score on a scale
  Change at Week 6 | -0.4 [-1.1 to 0.3] | 0.3 [-0.6 to 1.2]
  Change at Week 12: number analyzed (Participants) | 28 | 12
  Change at Week 12 | -0.8 [-1.5 to -0.1] | -0.1 [-1.1 to 0.8]

10. Secondary Outcome: PROMIS Short Form (SF) v1.0 General Self-Efficacy 4a
Description: The PROMIS Short Form (SF) v1.0 General Self-Efficacy 4a consists of 4 items rated on a 5-point Likert scale (not at all confident (1) to very confident (5)); values range from 4-20. Higher scores indicate higher levels of general self-efficacy.
Time Frame: Change from Baseline to 6 weeks (primary end point), persisting at 12 weeks
Population: The control group had one participant who did not complete week 12 testing.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 28 | 13
score on a scale
  Change at Week 6 | -0.3 [-1.9 to 1.3] | -0.2 [-2.3 to 1.9]
  Change at Week 12: number analyzed (Participants) | 28 | 12
  Change at Week 12 | 0.1 [-1.5 to 1.7] | 0.2 [-1.9 to 2.3]

11. Secondary Outcome: PROMIS Short Form (SF) Self-Efficacy for Managing Chronic Conditions
Description: The PROMIS Short Form (SF) Self-Efficacy for Managing Chronic Conditions is an 8-item scale rated on a 5-point Likert scale;values range from 8-32. Higher scores indicate higher levels of self confidence in one's ability to successfully perform specific tasks or behaviors related to one's health in a variety of situations.
Time Frame: Change from Baseline to 6 weeks (primary end point), persisting at 12 weeks
Population: The control group had one participant who did not complete week 12 testing.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 28 | 13
score on a scale
  Change at Week 6 | 2.2 [-1.4 to 5.8] | 2.7 [-2.0 to 7.5]
  Change at Week 12: number analyzed (Participants) | 28 | 12
  Change at Week 12 | 3.9 [0.2 to 7.5] | 4.4 [-0.4 to 9.2]

12. Secondary Outcome: PROMIS Scale v1.2 Global Health:
Description: The PROMIS Scale v1.2 Global Health measures quality of life on two domains: physical and mental health. Raw values for each domain range from 4 - 20; scores are converted to a t-score with a mean of 50 and SD of 10. Higher scores indicate better health.
Time Frame: Change from Baseline to 6 weeks (primary end point), persisting at 12 weeks
Population: The control group had one participant who did not complete week 12 testing.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 28 | 13
score on a scale
  Change at Week 6 | 0.5 [-2.8 to 3.8] | 2.1 [-2.3 to 6.5]
  Change at Week 12: number analyzed (Participants) | 28 | 12
  Change at Week 12 | 3.0 [-0.3 to 6.3] | 4.6 [0.1 to 9.0]

13. Secondary Outcome: Montreal Cognitive Assessment (MoCA)-BLIND
Description: The MoCA-BLIND assesses different cognitive domains: attention, concentration, memory, language, conceptual thinking, calculations, and orientation. The MoCA-BLIND has removed assessments requiring vision, thus can be completed using telehealth or telephone assessments. Score range: 0-22, with 18-22 normal range.
Time Frame: Change from Baseline to week 12
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 28 | 12
score on a scale | 1.1 [0.3 to 2.0] | 0.5 [-0.7 to 1.6]

14. Secondary Outcome: Clinical Frailty Scale
Description: The Clinical Frailty scale is a self-report scale to estimate function. The participant selects perceived level of function prior to and following admission ranging from very active to bedridden/terminal. Score range: 1 (very fit) - 9 (terminally ill), with higher scores indicating higher levels of frailty.
Time Frame: Change from Baseline to 6 weeks (primary end point), persisting at 12 weeks
Population: The control group had one participant who did not complete week 12 testing.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 28 | 13
score on a scale
  Change at Week 6 | -0.5 [-0.8 to -0.1] | -0.4 [-0.9 to 0.2]
  Change at Week 12: number analyzed (Participants) | 28 | 12
  Change at Week 12 | -0.8 [-1.2 to -0.4] | -0.7 [-1.2 to -0.2]

15. Secondary Outcome: Average Daily Step Count
Description: Average Daily Step Count per week will be collected via a Fitbit activity monitor. Higher step counts indicate higher level of physical activity.
Time Frame: Change from Baseline to 6 weeks (primary end point), persisting at 12 weeks
Population: One participant in the control group did not complete week 12.
Measure: Mean (95% Confidence Interval); unit: change in daily step count
Arm/Group | Intervention | Control
Number analyzed (Participants) | 27 | 13
change in daily step count
  Change at Week 6 | 56 [44 to 69] | 56 [44 to 69]
  Change at Week 12: number analyzed (Participants) | 27 | 12
  Change at Week 12 | 6 [-6 to 18] | 6 [-6 to 18]

16. Secondary Outcome: Patient Health Questionnaire 8 (PHQ8)
Description: The Patient Health Questionnaire 8 measures severity of depressive symptoms over the past 2 weeks. The 8 item scale is rated on a 4 point scale (not at all to nearly every day). Score range: 0-24. Higher scores indicate more severe depressive symptoms.
Time Frame: Change from Baseline to 6 weeks (primary end point), persisting at 12 weeks
Population: The control group had one participant who did not complete week 12 testing.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 28 | 13
score on a scale
  Change at Week 6 | -3.8 [-5.8 to -1.8] | -1.9 [-4.4 to 0.6]
  Change at Week 12: number analyzed (Participants) | 28 | 12
  Change at Week 12 | -5.0 [-7.0 to -2.9] | -3.1 [-5.6 to -0.5]

ADVERSE EVENTS:
Time Frame: 12 Weeks
Description: All safety events were categorized and counted and falls were graded according to the Falls-Grading Scale.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/15
Serious Adverse Events (participants affected / at risk) | 2/29 | 1/15
Other Adverse Events (participants affected / at risk) | 0/29 | 6/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=29) | Control (N=15)
Hospitalization (General disorders) | 2 (2) | 1 (1) — 2 participants were hospitalized for shortness of breath. 1 participant was hospitalized after being found passed out.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=29) | Control (N=15)
Falls (Injury, poisoning and procedural complications) | 0 (0) | 6 (8) — Falls were graded according to the Falls-Grading Scale.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-05): https://cdn.clinicaltrials.gov/large-docs/45/NCT04663945/Prot_SAP_000.pdf
  • Informed Consent Form (2022-05-05): https://cdn.clinicaltrials.gov/large-docs/45/NCT04663945/ICF_001.pdf